CLINICAL TRIAL: NCT01231893
Title: Transplantation of Autologous Olfactory Ensheathing Cells for Treatment of Complete Human Spinal Cord Injuries- a Phase I Clinical Trial.
Brief Title: Transplantation of Autologous Olfactory Ensheathing Cells in Complete Human Spinal Cord Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wroclaw Medical University (Other)
Collaborators: Institute of Immunology and Experimental Therapy of the Polish Academy of Sciences (Other); Department of Rehabilitation in Spinal Cord Injuries Akson (Unknown)
Responsible Party: Prof. Wlodzimierz Jarmundowicz, Department of Neurosurgery of the Wroclaw Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SR 406
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Complete Spinal Cord Injuries
Keywords: human, spinal cord injury, olfactory ensheathing cells, transplantation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- olfactory ensheathing cell recipient (Experimental)
  Interventions: Procedure: olfactory mucosa ensheathing cell grafting, rehabilitation
- control (Active Comparator)
  Interventions: Other: rehabilitation

INTERVENTIONS:
Procedure: olfactory mucosa ensheathing cell grafting, rehabilitation — In this group patients are planned to underwent a biopsy of their own olfactory mucosa for isolation and culture of olfactory ensheathing cells and olfactory fibroblasts. The suspension of these cells will be next transplanted into the focus of spinal cord injury. Before and after surgery the patients will undergo an intense neurorehabilitation program.
  Arms: olfactory ensheathing cell recipient
Other: rehabilitation — In this group the patients will not undergo any surgical procedure. They will participate in the same rehabilitation protocol that is planned for the patients from the experimental group.
  Arms: control

SUMMARY:
The purpose of this experimental therapy is an assessment of the safety and feasibility of transplantation of autologous olfactory ensheathing glia and olfactory fibroblasts obtained from the olfactory mucosa in patients with complete spinal cord injury.

DETAILED DESCRIPTION:
The increasing number of patients (mostly young), who have sustained a spinal cord injury mainly as a result of motor vehicle accidents, falls or violence has become worldwide a serious clinical, social and economical problem. Most accepted treatment protocols for spinal cord injury focus on techniques of early neuro-protection aimed at maximal prevention of secondary spinal cord injury (administration of methylprednisolon and spinal cord surgical decompression) as well as on methods of stimulation of plasticity in the central nervous system (neurorehabilitation). While these methods have been shown to stimulate functional recovery in patients with incomplete spinal cord injury, the results of treatment of patients with severe incomplete and complete spinal cord injuries remain unsatisfactory. This is due to the lack of spontaneous regeneration of lesioned axons in the spinal cord. Results from a substantial number of animal experiments performed mainly on the model of mammalian spinal cord injury in the last 3 decades led to the establishment of numerous regeneration-promoting strategies including application of neurotrophic factors, antibodies blocking the myelin-associated proteins and transplantation of cells with neurotrophic activity. Olfactory ensheathing cells (OECs) are an unique population of macroglia found in the lamina propria of olfactory mucosa, around the olfactory nerve fascicles and in the two outer layers of the olfactory bulb. These cells have the natural ability to stimulate the regrowth of lesioned peripheral and central axons. In a Phase I non-randomized controlled prospective study we have tested the hypothesis that a combined approach for treatment of complete spinal cord injuries consisting of intraspinal transplantation of a mixture of autologous OECs and fibroblasts isolated from the olfactory mucosa, combined with intense neuro-rehabilitation is safe and feasible.

ELIGIBILITY:
Inclusion Criteria:

* spinal cord injury at subacute or chronic stage
* a single spinal cord injury between segments C5 and L5
* myelopathy confirmed by MRI, not exceeding 2 spinal cord segments
* loss of sensory and motor function below the injury, confirmed in control studies (ASIA Category A)
* age from 16 to 65 years
* patient undergoing continuous rehabilitation
* good patient motivation and cooperation
* signed informed consent

Exclusion Criteria:

* a coexisting lesion of the nervous system
* progressive post-traumatic syringomyelia
* significant spinal stenosis or instability
* persistent neuropathic pain
* muscle atrophy or joint ossifications
* severe systemic disease (neoplasm, contagious disease, diabetes etc.)
* chronic sinusitis
* tumors or polyps of nasal cavities
* persistent hyposmia or anosmia
* pregnant or breastfeeding women

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-05

CONTACTS AND LOCATIONS:
Overall Officials: Wlodzimierz Jarmundowicz, M.D. Ph.D., Study Director — Department of Neurosurgery of Wroclaw Medical University; Pawel Tabakow, M.D. Ph.D., Principal Investigator — Department of Neurosurgery of Wroclaw Medical University
Locations (1):
- Department of Neurosurgery of Wroclaw Medical University, Wroclaw, Poland

REFERENCES:
- See also: Related Info — http://www.sci-therapies.info